CLINICAL TRIAL: NCT07358936
Title: THE EFFECTS OF CORRECTIVE EXERCISE AND KİNESİOTAPE APPLICATIONS ON PERFORMANCE AND FUNCTIONAL MOBILITY IN YOUNG BASKETBALL PLAYERS
Brief Title: THE EFFECTS OF CORRECTIVE EXERCISE AND KT APPLICATIONS IN YOUNG BASKETBALL PLAYERS
Acronym: KT:KINESIOTAPE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vedat Göken (Other)
Responsible Party: Sponsor-Investigator, Vedat Göken, Asistant Professor, Istinye University
Organization: Istinye University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 25-112
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Youth; Sport Performance
Keywords: YOUNG BASKETBALL PLAYERS; Corrective Exercise; Kinesiotape; Sport Performance
MeSH Terms: interventions — Athletic Tape

STUDY DESIGN:
Intervention Model Description: The athletes in the study will be divided into 3 groups. The first group will not receive any intervention and will continue their routine training. The second group will perform corrective exercises twice a week and will continue their routine training. The third group will continue their routine training along with kinesio taping twice a week.
  Kinesio Taping (KT) Application: This is a drug-free elastic band application applied to the muscle to reduce pain, increase circulation, provide muscle support, and improve joint stability.
  Corrective Exercise Program: These are exercises given to correct impaired movement patterns and improve posture. With these exercises, the quality of movement increases, the risk of injury decreases, and functional performance improves. Based on the athlete's initial assessment, a personalized exercise program will be designed for the athlete using artificial intelligence via a functional movement scanning system.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Corrective Exercise Group (Active Comparator): Based on the athlete's initial assessment, in addition to routine training, a personalized exercise program will be designed for the athlete using artificial intelligence via a functional movement scanning system; this will be performed twice a week for 6 weeks.
  Interventions: Procedure: Corrective Exercise
- Kinesiotape Group (Active Comparator): Based on the athlete's initial assessment, in addition to routine training, kinesio taping was applied to the deltoid muscle and quadriceps femoris muscle twice a week for 6 weeks.
  Interventions: Procedure: Kinesiotape
- Control Group (No Intervention): After the initial assessment, the athletes continued their routine training for 6 weeks.

INTERVENTIONS:
Procedure: Kinesiotape — This is a drug-free elastic band application applied to the muscle to reduce pain, increase circulation, provide muscle support, and improve joint stability.
  Arms: Kinesiotape Group
Procedure: Corrective Exercise — These exercises are given to correct disrupted movement patterns and improve posture.
  Arms: Corrective Exercise Group

SUMMARY:
The main objective of this research is to comparatively examine the effects of corrective exercise programs and kinesio taping (KT) applications on performance parameters and functional mobility in adolescent male basketball players. Kinesio taping is used with the aims of regulating muscle tone, increasing proprioception, improving circulation, and supporting pain management. In this context, corrective exercises are applied to correct movement disorders, eliminate musculoskeletal imbalances, and improve the functional movement quality in athletes. Although the effects of both methods on the performance parameters and functional mobility of athletes have been examined separately in the literature, a direct comparative study in adolescent basketball players is noticeable.

DETAILED DESCRIPTION:
Basketball is characterized by dynamic movement patterns involving high intensity, multi-plane, and sudden changes in direction. These characteristics require athletes to have highly developed physical parameters such as balance, strength, flexibility, and coordination. At the same time, the application of supportive methods to minimize the risk of injury without experiencing performance loss is of great importance in terms of training science and athlete health.

This research aims to achieve the following objectives:

Comparison of the effects of corrective exercise and chemotherapy on functional mobility in young basketball players, Analysis of the effects of both methods on fundamental performance parameters such as vertical jump, balance, acceleration, and change of direction, Measurement of pre- and post-application improvement levels through functional movement screening tests (e.g., Y-balance test, single-leg squat test, overhead squat, etc.), Evaluation of the effect of chemotherapy when combined with a corrective exercise program compared to applications performed alone, Providing concrete suggestions that can be used in planning preventive and performance-enhancing approaches for young basketball players. This research contains measurable objectives based on scientific data and is applicable in a short time, and aims to obtain important findings that will contribute to the performance development of young athletes in the field of sports science.

The study will include a total of 45 basketball players from Avrupa Karşıyaka Sports Club. The players will be divided into three groups using a simple lottery method: a kinesio taping group, a corrective exercise group, and a control group. Study timeline: The project will be completed within 12 months after obtaining ethical approval from the İstinye University Human Research Ethics Committee.

Sample and research group: Basketball players from Avrupa Karşıyaka Sports Club will be included in the study. 45 volunteer players meeting the inclusion criteria will be included. The sample size was calculated using *Power Version 3.1 software. For our study, with 80% power and a type 1 error of 0.05, and a moderate effect size (effect size = 0.54), it was found that a total of 45 people should be included in the study, with 15 people in each of the three different groups, to compare the effects.

ELIGIBILITY:
Inclusion Criteria:

* The male athlete's sport must be basketball.
* The male athlete must be between 9 and 16 years old.

Exclusion Criteria:

* Having undergone any surgical operation within the last 6 months.
* Having suffered a lower/upper extremity injury within the last 3 months.
* The volunteer does not wish to continue the study.
* Athletes for whom the necessary assessments or procedures could not be performed were excluded.

Ages: 9 Years to 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-05-16 (Estimated)

PRIMARY OUTCOMES:
Y Balance Test | From enrollment to the end of treatment at 3 weeks and 6 weeks
  The Y Balance Test is a widely used test in clinics and sports performance centers to assess dynamic balance in athletes. The test consists of a support platform with three PVC tubes attached in anterior, posteromedial, and posterolateral directions. The rear tubes are positioned at a 135-degree angle to the front tube, with a 45-degree angle between them. Each tube is marked at 5-millimeter intervals for measurement purposes.
  During the test, the support foot is held in the center of the measurement mechanism, while the other foot pushes against targets in the anterior, posteromedial, and posterolateral reach directions of the system using the toes, without losing balance or stepping on the targets. The aim is to measure the longest distance the target can reach.
Functional Movement System(FMS) | From enrollment to the end of treatment at 3 weeks and 6 weeks
  Used in athletes to identify movement patterns, mobility and stability deficiencies, and to predict injury risk. FMA is a test battery that evaluates individuals in terms of dynamic and functional capacity, essentially aiming to assess basic movement performance. The exercises in the Functional Movement Assessment allow for the identification of asymmetries, limitations, and compensations not only at the joint level but also throughout the movement pattern, thus enabling the early prediction and prevention of injury risk during physical activity. The test consists of seven movements: deep squat, high step, cross step, shoulder mobility, active straight leg raise, trunk stability, and rotational stability. Separate scoring is provided for each side in some movements, and athletes can receive a score between 0 and 21 on this test. If the test score is below 14, it suggests a potential risk of injury and a decrease in functional mobility capacity. Each movement should be repeated at leas
Agility T test | From enrollment to the end of treatment at 3 weeks and 6 weeks
  This is a test that evaluates an athlete's agility, speed, sudden changes of direction, balance, and coordination. Agility is defined as the ability to move the body between two points and change direction as easily, quickly, fluidly, and controllably as possible, along with balance, speed, strength, and neuromuscular coordination. Agility is considered a significant determining factor affecting performance, especially in team sports such as basketball. Previous studies have indicated that when developing agility skills, it is more accurate to evaluate it as a kinetic chain function involving the active participation of the entire body, rather than focusing solely on the muscles of the lower extremities.
My Jump 2 | From enrollment to the end of treatment at 3 weeks and 6 weeks
  This test, performed using a mobile application, assesses lower extremity strength and performance by calculating the athlete's jump height and flight time. In recent years, with advancements in technology, mobile applications aimed at improving, measuring, and analyzing athletic performance have continued to develop. One such application, My Jump 2, allows for a practical and rapid assessment of jump performance. The application aims to provide accurate calculations by considering flight time based on takeoff and landing frames. Since its introduction to the literature, the test has been used in numerous scientific studies.
Seated Medicine Ball Throw Test | From enrollment to the end of treatment at 3 weeks and 6 weeks
  This is a test used to measure an athlete's upper extremity strength. It is frequently used because it is easy to administer and inexpensive. Also known as the Medicine Ball Throw Test, it is a field test applied to evaluate upper extremity strength before and after training. There are various methods for evaluating upper extremity muscle strength. Compared to other tests, the Seated Medicine Ball Throw Test is frequently preferred due to its ease of application, cost, physical requirements, and practicality. In the SMBT test, the individual throws a shuttle ball as far as possible from a fixed seated position, and the test administrator measures the distance from the starting point of the throw to the point where the ball first touches the ground.
The Closed Kinetic Chain Lower Extremity Stability Test | From enrollment to the end of treatment at 3 weeks and 6 weeks
  It is a test designed to assess balance and endurance, evaluating an athlete's stability in a closed kinetic chain position. It provides performance-based, quantitative data aimed at assessing lower extremity stability within a closed kinetic chain context.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Istinye University, Istanbul, Istanbul
  - Istinye University, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided
I haven't decided yet.